CLINICAL TRIAL: NCT03743805
Title: Rapid Reversal of CNS-Depressant Drug Effect Prior to Brain Death Determination
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Insufficient patients
Sponsor: Prisma Health-Midlands (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00077995
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Brain Death; Anoxic Brain Injury; Cardiac Arrest; Sedative Intoxication; Narcotic Intoxication
Keywords: brain; death; sedative; narcotic
MeSH Terms: conditions — Brain Death; Hypoxia-Ischemia, Brain; Heart Arrest; Death | interventions — Flumazenil; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Reversal drugs (Experimental): Flumazenil and naloxone
  Interventions: Drug: Flumazenil; Drug: Naloxone

INTERVENTIONS:
Drug: Flumazenil — 0.2 mg IV push, which may be repeated every 20 minutes for up to a total of 1 mg
  Other Names: Romazicon
Drug: Naloxone — 0.4 mg IV push, which may be repeated every 2 minutes for up to a total of 2 mg
  Other Names: Narcan; Evzio

SUMMARY:
Current standard of care prior to determination of brain death in subjects with suspected anoxic brain injury is to exclude complicating medical conditions that may confound clinical assessment (such as severe electrolyte, acid base, endocrine or circulatory disturbance), achieve normothermia and normal systolic blood pressure over 100 mmHg (with or without vasopressor use), exclude the presence of neuromuscular blocking agents (with the presence of a train of 4 twitches with maximal ulnar nerve stimulation) as well as to exclude the presence of CNS depressant drug effects. At the present time the latter is done by history, drug screen and allowing enough time for paralytic and sedative drugs to be metabolized and cleared from the body. Clearance is calculated by using 5 times the drug's half-life assuming normal hepatic and renal functions. Half-life can also be prolonged in subjects who have been treated with induced hypothermia. Literature search revealed articles with general guidelines and approaches to brain death, but none addressed pharmacological reversal of sedative drugs

DETAILED DESCRIPTION:
Question of proposed study is whether a subject's comatose state is secondary to delayed clearance of a previously administered CNS depressant. By using pharmacologic reversal agents of commonly used benzodiazepines and opioids, the investigators aim to identify participants that may likely improve after complete clearance of the drugs from their system.

Prospective trial with enrollment of 30 subjects in 2 intensive care units at Palmetto Health Richland from January 1st 2019 to June 30th 2020. Research procedures will be performed in the intensive care setting. If participants had undergone targeted temperature management (33-36 degrees Celsius for 24 hours via intravascular or surface control methods, with or without sedation or neuromuscular blockade, followed by rewarming actively or passively at 0.25-0.5 degrees per hour over 8-12 hours to 37 degrees) investigators will wait 24 hours after rewarming prior to testing. End point is to evaluate if pharmacological reversal agents would result in improved GCS scores or return of cerebral or brainstem functions in some comatose subjects, which will be considered a positive test result.

ELIGIBILITY:
Inclusion Criteria:

* Adults with cardiac arrest who may have completed targeted temperature management (hypothermia protocol) and have had no neurological recovery after 24 hours of rewarming will be enrolled. Subjects will have a suspected diagnosis of anoxic brain injury secondary to cardiac arrest, and seizures ruled out with an EEG. All subjects are expected to be unable to consent and consent will be obtained from their legal authorized representative.

Exclusion Criteria:

* Spontaneous recovery of neurological functions, presence of seizures on EEG, individuals who are not yet adults, pregnant women and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Improved GCS scores or return of cerebral or brainstem functions in comatosed subjects | Within 30 minutes post treatment
  Subjects will be observed closely and tested before and after intervention for any signs of cerebral or brainstem function (1-Response to pain stimulus with earlobe pinching, trapezius squeezing and sternal rub or other brain-originating movements, e.g. seizures, decerebrate or decorticate posturing. 2-Pupillary light reflex with bright light. 3-Corneal reflexes with the use of cotton swab or tissue paper. 4-Gag reflex with a tongue depressor looking for bilateral palatal elevation. 5-Cough with tracheal suctioning at the carinal level) and GCS re-evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Sameh R Hanna, MD, Principal Investigator — Palmetto Health-University of South Carolina Medical Group
Locations (1):
- PRISMA Health Midlands, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Varelas PN, Lewis A. Modern Approach to Brain Death. Semin Neurol. 2016 Dec;36(6):625-630. doi: 10.1055/s-0036-1592317. Epub 2016 Dec 1. PMID 27907967
- [Background] Wijdicks EF. Brain death guidelines explained. Semin Neurol. 2015 Apr;35(2):105-15. doi: 10.1055/s-0035-1547532. Epub 2015 Apr 3. PMID 25839719
- [Background] Gardiner D, Shemie S, Manara A, Opdam H. International perspective on the diagnosis of death. Br J Anaesth. 2012 Jan;108 Suppl 1:i14-28. doi: 10.1093/bja/aer397. PMID 22194427
- [Background] Wijdicks EF. Brain death worldwide: accepted fact but no global consensus in diagnostic criteria. Neurology. 2002 Jan 8;58(1):20-5. doi: 10.1212/wnl.58.1.20. PMID 11781400
- [Background] Wijdicks EF. The diagnosis of brain death. N Engl J Med. 2001 Apr 19;344(16):1215-21. doi: 10.1056/NEJM200104193441606. No abstract available. PMID 11309637
- [Background] Wijdicks EF. Determining brain death in adults [RETIRED]. Neurology. 1995 May;45(5):1003-11. doi: 10.1212/wnl.45.5.1003. No abstract available. PMID 7746373
- [Background] Wahlster S, Wijdicks EF, Patel PV, Greer DM, Hemphill JC 3rd, Carone M, Mateen FJ. Brain death declaration: Practices and perceptions worldwide. Neurology. 2015 May 5;84(18):1870-9. doi: 10.1212/WNL.0000000000001540. Epub 2015 Apr 8. PMID 25854866
- [Background] Wijdicks EF, Varelas PN, Gronseth GS, Greer DM; American Academy of Neurology. Evidence-based guideline update: determining brain death in adults: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2010 Jun 8;74(23):1911-8. doi: 10.1212/WNL.0b013e3181e242a8. PMID 20530327
- [Background] Greer DM, Varelas PN, Haque S, Wijdicks EF. Variability of brain death determination guidelines in leading US neurologic institutions. Neurology. 2008 Jan 22;70(4):284-9. doi: 10.1212/01.wnl.0000296278.59487.c2. Epub 2007 Dec 12. PMID 18077794
- [Background] Shappell CN, Frank JI, Husari K, Sanchez M, Goldenberg F, Ardelt A. Practice variability in brain death determination: a call to action. Neurology. 2013 Dec 3;81(23):2009-14. doi: 10.1212/01.wnl.0000436938.70528.4a. Epub 2013 Nov 6. PMID 24198290